CLINICAL TRIAL: NCT07034040
Title: SmaRTWork - a Decision Support System to Promote Return to Work Among People Sick-listed With Musculoskeletal Disorders
Acronym: SmaRTWork
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 563919; 315041 (Other Grant/Funding Number: The Research Council of Norway)
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Sick Leave; Musculoskeletal
Keywords: Sick leave; musculoskeletal disorder; sickness absence; return to work; mHealth
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SmaRTWork (Experimental): This group receives the SmaRTWork intervention in addition to usual care
  Interventions: Behavioral: SmaRTWork
- Usual care (No Intervention): The participants receive usual care as if they were not part of any study. There are no restrictions on what they can or cannot do.

INTERVENTIONS:
Behavioral: SmaRTWork — The SmaRTWork app provides weekly individually tailored self-management plans by matching the participant's health information and sick leave status with targeted educational messages, physical activity advice, and exercise recommendations. In addition, participants with specific problems regarding i) work accommodations, ii) workplace conflicts, iii) large responsibilities as caregivers, iv) financial problems, or v) who do not think they will return to the old workplace are offered to be set in contact with a caseworker at the social insurance office. The intervention is given in addition to usual care.
  Arms: SmaRTWork

SUMMARY:
The objective of this study is to evaluate the effect of an intervention, SmaRTWork, on return to work compared to usual care for individuals who are sick-listed due to musculoskeletal disorders. Potential participants are individuals of working age (20-59 years) sick-listed due to a musculoskeletal disorder (neck pain, low back pain, or widespread pain) for up to 12 weeks living in Norway. The primary outcome will be time to sustainable return to work. We will also evaluate the effect on other work outcomes and health outcomes. We will also interview participants and stakeholders about their experience with the intervention.

DETAILED DESCRIPTION:
The objective of this study is to determine the effectiveness of SmaRTWork (intervention) on return to work (RTW) compared to usual care (comparator) for individuals sick-listed due to musculoskeletal disorders. The study is designed as a single-blinded randomised controlled trial (RCT) with two parallel groups. Individuals of working age (20-59 years) sick-listed due to a musculoskeletal disorder (neck pain, low back pain, or widespread pain) for up to 12 weeks living in Norway are eligible for the study. Potential participants are identified and informed about the project by their general practitioner. We plan to include a total of 298 participants in the trial (and 15-20 in a pilot, giving a total of 318). The primary outcome will be time to sustainable RTW, i.e., one month without receiving sickness benefits, during the 12 months of follow-up based on registry data. Secondary outcomes include other work outcomes and health outcomes. Along with the RCT we will also conduct qualitative studies and a process evaluation. If the SmaRTWork turns out to be effective on RTW, we will also perform a health economic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 20-59 years old (working age)
* Living in Norway
* Sick-listed due to a musculoskeletal disorder for up to 12 weeks
* Musculoskeletal complaints are the main reason for sick leave.
* The main diagnosis for sick leave is unspecific pain, for example one of the following (ICPC-2 diagnoses codes):
* Neck symptom/complaint (L01)
* Back symptom/complaint (L02)
* Low back symptom/complaint (L03)
* Muscle pain (L18)
* Back syndrome without radiating pain (L84)

Exclusion Criteria:

* Do not have a smartphone with internet access (i.e., to be able to download and access the SmaRTWork app).
* Pregnant
* No employer (unemployed or self-employed)
* Poor Norwegian comprehension
* Sick listed for more than 3 months the last year
* Have a planned date for RTW during the next week
* Have previously participated in the study or currently participating in other studies
* Unable to take part in exercise/physical activity (e.g., use of walking aids, unable to get up and down on the floor independently)
* Leg pain worse than back pain
* Red flags that could indicate serious underlying pathology:

  * Changes in bladder or bowel function
  * General feeling of being unwell (malaise), fever and/or unexplained weight loss
  * Reduced muscle (motor) function, sensory loss, walking problems or balance problems
  * Neck or back pain that started after the age of 55 or feel different from previous pain episodes
  * Pain that does not improve with rest or light activity or pain that is much worse during the night
  * Previous or ongoing cancer
  * Use of steroids/immune suppressing medications or drug use
  * Pain that is trauma (injury) related
* Serious ongoing somatic (e.g., unstable heart disease) or mental disorder (e.g., psychosis, ongoing manic episode, suicidal ideation) that prevents participation
* Pain has not been assessed by a physician

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 298 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Time to sustainable return-to-work (RTW) | 12 months from randomization
  Time to sustainable return-to-work (RTW), i.e., one month without receiving sickness benefits, during the 12 months of follow-up from randomization based on registry data

SECONDARY OUTCOMES:
Number of sickness absence days | 12 months from randomization
  Total number of sickness absence days during 12 months of follow-up from randomization based on registry data
Probability of working each month | 12 months from randomization
  The probability of working (i.e., not receiving medical benefits) each month during 12 months of follow-up, measured as repeated events
Musculoskeletal Health Questionnaire (MSK-HQ) | From randomization to 12 months of follow-up
  Questionnaire that measures musculoskeletal health with scores from 0 to 56 points, with higher scores indicating better musculoskeletal health
Health-related quality of life | 12 months from randomization
  Assessed by the EuroQol 5-dimension questionnaire, weighted according to the Danish value set (range, 0-1, with higher scores indicating better health status) and the EuroQol visual analog scale (range, 0-100, with higher scores indicating better health status)
Average pain last week | 12 months from randomization
  Measured by a numeric rating scale scores from 0 (no pain) to 10 (worst imaginable pain)
Pain Self-Efficacy | 12 months from randomization
  Ability to cope despite pain as assessed with the Pain Self-Efficacy Questionnaire (PSEQ), range, 0-60, with higher scores indicating greater confidence
Depressive symptoms | 12 months from randomization
  Depressive symptoms by the Patient Health Questionnaire-2 (PHQ-2), scores range from 0-6 (higher more symptoms)
Brief Illness Perception | 12 months from randomization
  Cognitive and emotional perceptions of illness assessed by the Brief Illness Perception Questionnaire (range, 0-80, with higher scores indicating greater illness perception)
Work ability | 12 months from randomization
  Work ability measured by the single item from the Work Ability Index (WAI) scored from 0 (worst) to 10 (best).
Overall improvement | 12 months from randomization
  Assessed by the Global Perceived Effect scale. Range, -5 to 5, with positive scores indicating improvement of pain
Fear avoidance beliefs | 12 months from randomization
  Measured by one-item from Tampa Scale of Kinesiophobia scored from 0 (no fear) to 10 (much fear)

CONTACTS AND LOCATIONS:
Overall Officials: Lene Aasdahl, MD PhD, Principal Investigator — Norwegian University of Science and Technology; Solveig K Grudt, Head of Department, Study Chair — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No
Due to the ethical consent data cannot be shared.